CLINICAL TRIAL: NCT06108830
Title: Effect of Esketamine Combined With Remimazolam on Postoperative Sleep Disturbance and Anxiety in Patients Undergoing Gastroenteroscopies
Brief Title: Esketamine Combined With Remimazolam on Postoperative Sleep Disturbance and Anxiety in Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GWang024
Record Dates: First submitted 2023-08-27; First posted 2023-10-31 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Sleep Disturbance
Keywords: Esketamine; remimazolam; anxiety; gastroenteroscopy
MeSH Terms: conditions — Parasomnias; Anxiety Disorders | interventions — Esketamine; remimazolam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group of patients undergoing gastroenteroscopies with normal saline (Placebo Comparator): Patients undergoing gastroenteroscopies were given propofol 2-3mg/kg and 10ml 0.9% saline before the procedure began
  Interventions: Drug: normal saline
- Group of patients undergoing gastroenteroscopies with esketamine (Active Comparator): Patients undergoing gastroenteroscopies were given propofol 2 to 3mg/kg and esketamine 0.2mg/kg before the procedure began
  Interventions: Drug: Esketamine
- Group of patients undergoing gastroenteroscopies with remimazolam (Active Comparator): Patients undergoing gastroenteroscopies were given propofol 2 to 3mg/kg and remimazolam 0.15mg/kg before the procedure began
  Interventions: Drug: Remimazolam
- Group of patients undergoing gastroenteroscopies with remimazolam and esketamine (Active Comparator): Patients undergoing gastroenteroscopies were given propofol 2 to 3mg/kg， esketamine 0.2mg/kg and remimazolam 0.15mg/kg before the procedure began
  Interventions: Drug: Esketamine and remimazolam

INTERVENTIONS:
Drug: Esketamine — Patients undergoing gastroenteroscopies were given propofol 2 to 3mg/kg and esketamine 0.2mg/kg before the procedure began
  Other Names: Group of patients undergoing gastroenteroscopies with esketamine
  Arms: Group of patients undergoing gastroenteroscopies with esketamine
Drug: Remimazolam — Patients undergoing gastroenteroscopies were given propofol 2 to 3mg/kg and remimazolam 0.15mg/kg before the procedure began
  Other Names: Patients undergoing gastroenteroscopies were given propofol 2 to 3mg/kg and remimazolam 0.15mg/kg before the procedure began
  Arms: Group of patients undergoing gastroenteroscopies with remimazolam
Drug: Esketamine and remimazolam — Patients undergoing gastroenteroscopies were given propofol 2 to 3mg/kg and remimazolam 0.15mg/kg before the procedure began
  Other Names: Patients undergoing gastroenteroscopies were given propofol 2 to 3mg/kg， esketamine 0.2mg/kg and remimazolam 0.15mg/kg before the procedure began
  Arms: Group of patients undergoing gastroenteroscopies with remimazolam and esketamine
Drug: normal saline — Patients undergoing gastroenteroscopies were given propofol 2-3mg/kg and 10ml 0.9% saline before the procedure began
  Other Names: Group of patients undergoing gastroenteroscopies with normal saline
  Arms: Group of patients undergoing gastroenteroscopies with normal saline

SUMMARY:
To explore the effects of esketamine combined with remimazolam on postoperative sleep disturbance and anxiety in surgical patients undergoing gastroenteroscopies

DETAILED DESCRIPTION:
Postoperative sleep disturbance (PSD) occur in the form of sleep deprivation, circadian rhythm disturbance, and structural abnormalities, and have a high incidence in patients undergoing surgery. Postoperative sleep disorders can lead to postoperative delirium and cognitive dysfunction, aggravate postoperative acute pain, and delay postoperative recovery.

Benzodiazepines have a certain sedative hypnotic anti-anxiety effect, and remimazolam as a new benzodiazepine, its sedative hypnotic anti-anxiety effect is worthy of further exploration.Esketamine is an NMDA receptor antagonist with analgesic and sedative effects, and is widely used in clinical treatment of refractory depression. For patients undergoing surgery, in addition to sedation and analgesia, whether the intraoperative use of esketamine has positive effects on postoperative sleep disturbance and anxiety is worth exploring.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-65 years old;
2. ASA classification is grade I-III;
3. Elective surgery is proposed
4. BMI of 19-30 kg/m2;
5. Patients who agreed to enroll in this study voluntarily

Exclusion Criteria:

1. Those who are known to be allergic to the drug ingredients in this study and their allergic constitution;
2. Allergic history of general anesthesia drugs, opioid drugs, non-steroidal drugs;
3. History of neurological diseases; History of chronic pain; Drug and alcohol addiction; A long history of opioid use; Opiates were given 48 hours before surgery;
4. ASA rating of IV or V;
5. Coronary heart disease, bronchial asthma, severe hypertension, severe blood system dysfunction, liver and kidney function, electrolyte abnormalities;
6. History of gastrointestinal disease (peptic ulcer, Crohn's disease, ulcerative colitis);
7. Respiratory insufficiency, respiratory failure;
8. Patients who refused to use intravenous PCA for analgesia;
9. Pregnant or lactating women;
10. BMI<18 kg/m2 or BMI>30kg/m2;
11. Poor compliance, unable to complete the experiment according to the study plan;
12. Participants who have participated in clinical trials of other drugs within the last 4 weeks;
13. Any circumstances deemed unsuitable for inclusion by the researcher for any reason.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Sleep disturbance and anxiety after surgery | 1 day before surgery, 1 and 3 days after surgery
  Patients completed the sleep quality (AIS, Athens Insomnia Scale) and anxiety (Hospital Anxiety and Depression Scale) rating scales on the day before surgery. HADS consists of 14 items to calculate the patient's comprehensive score, including 7 anxiety related scores and 7 depression related scores. Each question in the questionnaire was scored on a scale of 0-3, so patients scored 0-21 on both anxiety and depression. Scores of 8 points or higher are diagnosed as depression or anxiety.And we asked the patients to fill out these questionnaires on the day 1 and 3 after surgery again to evaluate the changes in sleep quality and anxiety. (The AIS score ranges from 0 to 24 points, and a total score of 6 points or higher indicates a diagnosis of insomnia). . We recorded AIS scores, HDS-A scores and HDS-D scores as separate statistical indicators.

SECONDARY OUTCOMES:
Pain Score (NRS) | 1 and 3 days after surgery
  The pain score at rest or after movement was evaluated by pain 11-point numerical rating scale (NRS): 0 = no pain, 10 = greatest imaginable pain.
Incidence of injection pain | Intraoperative
  The frequency of injection pain induced by propofol was recorded
Dosage of drug | Intraoperative
  The dosage of propofol, esketamine and remimazolam were recorded
Mean intraoperative blood pressure | Intraoperative
  The mean intraoperative blood pressure was recorded
Oxygen saturation | Intraoperative
  The mean intraoperative oxygen saturation was recorded
Somatokinetic reaction | Intraoperative
  The number of intraoperative body movements was recorded
Operation time | Intraoperative
  The duration of the patient's operation was recorded(up to 24 h)
Duration of anesthesia | After surgery
  The patient's duration of anesthesia was recorded(up to 24 h)
Time of awakening | After surgery
  The duration from the end of anesthesia to recovery was recorded(up to 24 h)
Time to walking down | After surgery
  Record the time from waking up to walking down(up to 24 h)
Adverse event | Within 3 days after surgery
  All kinds of adverse events occurred in patients were recorded
Exhaust time | Within 3 days after surgery
  Records from end of anesthesia to patients with postoperative exhaust time for the first time

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, Study Director — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No